CLINICAL TRIAL: NCT03351335
Title: Open-label, Prospective Evaluation of the Ulthera® System for Lifting Submental (Under the Chin) and Neck Tissue in Chinese Patients
Acronym: ULT-302
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Collaborators: Ulthera, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M960001052
Record Dates: First submitted 2017-11-20; First posted 2017-11-22 (Actual); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2018-08

CONDITIONS: Mild to Moderate Skin Laxity Under the Chin; Mild to Moderate Skin Laxity on Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Ultherapy®, energy level 3 (Experimental): Group 1: Subjects will receive Ultherapy® treatment at energy level 3 (EL3).
  Interventions: Device: Microfocused ultrasound with visualization
- Ultherapy®, energy level 4 (Experimental): Group 2: Subjects will receive Ultherapy® treatment at energy level 4 (EL4).
  Interventions: Device: Microfocused ultrasound with visualization
- Ultherapy®, energy level 2 (Experimental): Group 3: Subjects will receive Ultherapy® treatment at energy level 2 (EL2).
  Interventions: Device: Microfocused ultrasound with visualization

INTERVENTIONS:
Device: Microfocused ultrasound with visualization — All subjects will receive an Ultherapy® treatment at dual depth using the 4-4.5mm and 7-3.0mm transducers. Treatments will be provided to the lower face, submental (under the chin) and neck area.
  Other Names: Ultherapy®

SUMMARY:
To evaluate the Ulthera® System for lifting submental (under the chin) and neck tissue in Chinese patients

ELIGIBILITY:
Inclusion Criteria:

1. Both parents of full Chinese decent.
2. Mild to moderate skin laxity of the submental (under the chin) and neck tissue as determined by the physician and trained assessors.
3. Adequate menton area to allow for quantitative analysis, as confirmed by photography images.
4. Willingness and ability to comply with protocol requirements, including returning for follow-up visit and abstaining from any other procedures in the areas to be treated through the follow-up period.
5. Subjects of childbearing potential must have a negative urine pregnancy test result and must not be lactating at the Screening Visit and be willing and able to use an acceptable method of birth control (e.g. barrier methods used with a spermicidal agent, hormonal methods, IUD, surgical sterilization, abstinence) during the study. Women will not be considered of childbearing potential if one of the following conditions is documented on the medical history:

   1. Postmenopausal with last menstrual bleeding at least 12 months prior to study; and
   2. Without a uterus and/or both ovaries.
6. Willing to take 600mg Ibuprofen as pre-treatment medication, at least 60 minutes but not more than two hours prior to study treatment.
7. Willingness and ability to provide written consent for study-required photography and adherence to photography procedures (i.e., removal of jewelry and makeup).
8. Willingness and ability to provide written informed consent prior to performance of any study-related procedure.

Exclusion Criteria:

1. Presence of an active systemic or local skin disease that may affect wound healing.
2. Presence of any hemorrhagic disorder or hemostatic dysfunction, herpes simplex, diabetes, epilepsy, bell's palsy or any physical or psychological condition that is deemed unacceptable by the investigator for participation in this study.
3. Severe solar elastosis.
4. Excessive subcutaneous fat in the area(s) to be treated.
5. Excessive skin laxity on the area(s) to be treated.
6. Significant scarring in the area(s) to be treated that would interfere with assessing results.
7. Open wounds or lesions in the area(s) to be treated.
8. Severe or cystic acne on the area(s) to be treated.
9. Active implants (e.g., pacemakers or defibrillators), or metallic implants in the treatment areas (dental implants not included.)
10. Inability to understand the protocol or to give informed consent.
11. Allergy or sensitivity to pre-treatment medication (ibuprofen).
12. Microdermabrasion, or prescription level glycolic acid treatment to the treatment area(s) within four weeks prior to study participation or during the study.
13. Marked asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring, or thick sebaceous skin in the area(s) to be treated.
14. BMI greater than or equal to 30.
15. History of chronic drug or alcohol abuse.
16. More than 2-3 doses of any NSAID in any 2-week period prior to and throughout study.
17. History of autoimmune disease.
18. Concurrent therapy that, in the investigator's opinion, would interfere with the evaluation of the safety or efficacy of the study device.
19. Subjects who anticipate the need for inpatient surgery or overnight hospitalization during the study.
20. Subjects who, in the investigator's opinion, have a history of poor cooperation, noncompliance with medical treatment, or unreliability.
21. Concurrent enrollment or enrollment in any study involving the use of investigational devices or drugs within the past three months.
22. Current smoker as defined by

    1. Having smoked one or more cigarettes per day on a daily basis within the past year; or
    2. Smoke cessation within the past 6 months.
23. Current user of any nicotine-containing products, e.g., e-cigarettes, Nicorette gum, nicotine patches, etc.
24. History of the following cosmetic treatments in the area(s) to be treated:

    1. Skin tightening procedure within the past year;
    2. Injectable filler of any type within the past: i) 9 months for Hyaluronic acid fillers (e.g. Restylane); ii) 24 months for Ca Hydroxyapatite fillers (e.g. Radiesse); iii) 12 months for Long-lasting Hyaluronic acid (Juvéderm Voluma); iv) 24 months for Poly-L-Lactic acid fillers (e.g. Sculptra); v) Ever for permanent fillers (e.g. Silicone, Artecoll)
    3. Neurotoxins within the past three months;
    4. Ablative resurfacing laser treatment;
    5. Nonablative, rejuvenative laser or light treatment within the past six months;
    6. Surgical dermabrasion or deep facial peels;
    7. Facelifts within the past year; or
    8. Any history of contour threads.
25. History (in the prior year) or current use of the following prescription medications:

    1. Accutane or other systemic retinoids within the past six months;
    2. Topical Retinoids within the past two weeks;
    3. Antiplatelet agents/Anticoagulants (Coumadin, Heparin, Plavix);
    4. Psychiatric drugs that in the investigators opinion would impair the subject from understanding the protocol requirements or understanding and signing the informed consent.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-08-10 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Kreymerman, MD, FA, Study Director — Merz North America, Inc.
Locations (7):
- United States (7):
  - Merz Investigational Site # 0010411, Los Gatos, California
  - Merz Investigational Site # 0010321, San Diego, California
  - Merz Investigational Site # 0010358, Vista, California
  - Merz Investigational Site # 0010410, Austin, Texas
  - Merz Investigational Site # 0010422, Bellaire, Texas
  - Merz Investigational Site # 0010423, Houston, Texas
  - Merz Investigational Site # 0010125, Plano, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 7 investigational sites in the United States.
Pre-assignment Details: A total of 180 participants were screened, out of which 60 were enrolled and treated. Of these, 56 participants completed the study.
Groups:
- Group EL 2: Ultherapy: Participants received a single Ultherapy treatment at energy level 2 (EL2) on the lower face, submental (under the chin) and neck area at dual depth using transducer DeepSEE (DS) 4 to 4.5 with treatment frequency 4 megahertz (MHz) and depth 4.5 millimeter (mm) at energy level 0.90 Joule (J), and transducer DS 7 to 3.0 with treatment frequency 7 MHz and depth 3.0 mm at energy level 0.30 J at baseline.
- Group EL 3: Ultherapy: Participants received a single Ultherapy treatment at energy level 3 (EL3) on the lower face, submental (under the chin) and neck area at dual depth using transducer DS 4 to 4.5 with treatment frequency 4 MHz and depth 4.5 mm at energy level 1.00 J and transducer DS 7 to 3.0 with treatment frequency 7 MHz and depth 3.0 mm at energy level 0.35 J at baseline.
- Group EL 4: Ultherapy: Participants received a single Ultherapy treatment at energy level 4 (EL4) on the lower face, submental (under the chin) and neck area at dual depth using transducer DS 4 to 4.5 with treatment frequency 4 MHz and depth 4.5 mm at energy level 1.20 J and transducer DS 7 to 3.0 with treatment frequency 7 MHz, and depth 3.0 mm at energy level 0.45 J at baseline.
Period: Overall Study
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Started | 21 | 19 | 20
Completed | 21 | 19 | 16
Not Completed | 0 | 0 | 4
Not completed — Failure to maintain inclusion/exclusion | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Population: The safety evaluation set (SES) population included all participants who were treated.
Groups:
- Group EL 2: Ultherapy: Participants received a single Ultherapy treatment at EL2 on the lower face, submental (under the chin) and neck area at dual depth using transducer DS 4 to 4.5 with treatment frequency 4 MHz and depth 4.5 mm at energy level 0.90 J, and transducer DS 7 to 3.0 with treatment frequency 7 MHz and depth 3.0 mm at energy level 0.30 J at baseline.
- Group EL 3: Ultherapy: Participants received a single Ultherapy treatment at EL3 on the lower face, submental (under the chin) and neck area at dual depth using transducer DS 4 to 4.5 with treatment frequency 4 MHz and depth 4.5 mm at energy level 1.00 J and transducer DS 7 to 3.0 with treatment frequency 7 MHz and depth 3.0 mm at energy level 0.35 J at baseline.
- Group EL 4: Ultherapy: Participants received a single Ultherapy treatment at EL4 on the lower face, submental (under the chin) and neck area at dual depth using transducer DS 4 to 4.5 with treatment frequency 4 MHz and depth 4.5 mm at energy level 1.20 J and transducer DS 7 to 3.0 with treatment frequency 7 MHz, and depth 3.0 mm at energy level 0.45 J at baseline.
- Total: Total of all reporting groups
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy | Total
Number analyzed (Participants) | 21 | 19 | 20 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.7 (6.4) | 49.4 (8.0) | 51.4 (7.2) | 52.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 17 | 18 | 56
  Male | 0 | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 21 | 19 | 20 | 60
Fitzpatrick skin type [Count of Participants; unit: Participants] — Skin type I = white; very fair, red or blonde hair blue eyes; freckles; always burns, never tans, skin type II = white, fair, red or blond hair; blue, hazel or green eyes; usually burns, tans with difficulty, skin type III = cream white; fair with any eye or hair color (common); sometimes mild burn, gradually tans, skin type IV = brown; typical Mediterranean Caucasian skin; rarely burns, tans with ease, skin type V = dark brown; mid-eastern skin types; very rarely burns, tans easily, and skin type VI = black; never burns, tans very easily.
  Participants
    Type I | 0 | 0 | 0 | 0
    Type II | 0 | 3 | 0 | 3
    Type III | 3 | 6 | 10 | 19
    Type IV | 15 | 8 | 9 | 32
    Type V | 3 | 1 | 1 | 5
    Type VI | 0 | 0 | 0 | 0
    Missing | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Overall Lifting and Tightening of Submental (Under the Chin) and Neck Tissue Area at Day 90 Post-treatment
Description: Lifting was determined by a quantitative measure of tissue lift in the area using photographs taken with Mirror Photofile software and a Vectra 3 dimensional (3D) digital imaging system. Mean change was calculated as mean of left and right side 90 day area minus mean of left and right baseline area.
Time Frame: Baseline and Day 90
Population: The full analysis set (FAS) population consisted of all participants in the SES population for whom the primary efficacy variable was available (that is all participants who had the baseline and post-baseline value of the primary efficacy variable).
Measure: Mean (Standard Deviation); unit: square millimeter (mm^2)
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Number analyzed (Participants) | 21 | 19 | 16
square millimeter (mm^2) | -14.4 (28.0) | -7.9 (40.8) | -22.3 (38.2)

2. Secondary Outcome: Number of Participants With Improvement From Baseline in Overall Lifting and Tightening of Submental (Under the Chin) and Neck Tissue Area as Assessed by Physician Global Aesthetic Improvement Scale (PGAIS) Scores at Day 90 Post-treatment
Description: Overall aesthetic improvement was assessed by a principal investigator using global aesthetic improvement scale (GAIS).The PGAIS was a 5-point scale (-2 to 2) that rates global aesthetic improvement from the pre-treatment appearance in which live observation and photo review were utilized by the physician. The ratings are -2 (much worse), -1 (worse), 0 (no change), 1 (improved), and 2 (much improved). Improvement was determined by participant response rate (improved or much improved) on PGAIS.
Time Frame: Day 90
Population: The FAS population consisted of all participants in the SES population for whom the primary efficacy variable was available (that is all participants who had the baseline and post-baseline value of the primary efficacy variable).
Measure: Count of Participants; unit: Participants
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Number analyzed (Participants) | 21 | 19 | 16
Participants | 18 | 16 | 16

3. Secondary Outcome: Number of Participants With Improvement From Baseline in Overall Lifting and Tightening of Submental (Under the Chin) and Neck Tissue Area as Assessed by Subject Global Aesthetic Improvement Scale (SGAIS) at Day 90 Post-treatment
Description: Overall aesthetic improvement was assessed by a principal investigator using GAIS. The SGAIS was a 5-point scale (-2 to 2) that rates global aesthetic improvement from the pre-treatment appearance in which live observation and photo review were utilized by the participant. The ratings are -2 (much worse), -1 (worse), 0 (no change), 1 (improved), and 2 (much improved). Improvement is determined by participant response rate (improved or much improved) on SGAIS.
Time Frame: Day 90
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Number analyzed (Participants) | 21 | 19 | 16
Participants | 17 | 14 | 16

4. Secondary Outcome: Number of Participants With Improvement From Baseline in Overall Lifting and Tightening of Submental (Under the Chin) and Neck Tissue Area as Assessed by a Masked, Qualitative Assessment of Photographs at Day 90 Post-treatment
Description: Masked, qualitative photographic assessment of photographs were obtained using Mirror Photofile software and a Vectra 3D digital imaging system. Experienced physicians evaluated paired pre- and 90-days post-treatment photographs of evaluable participants in a blinded fashion. Each blinded assessor reviewed the image sets and identified the post-treatment photographs according to the following definitions: Change (A change that is noticeable) and No Change (No change is apparent). Blinded assessors were asked to compare pre- and post-treatment photos for noticeable change. When change was noted the assessors were asked to determine which image demonstrated improvement. Assessor data were compiled and analyzed using majority rule for each participant assessed.
Time Frame: Day 90
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Number analyzed (Participants) | 21 | 19 | 16
Participants
  Improved: Left Side | 8 | 8 | 8
  Improved: Right Side | 10 | 9 | 8
  Improved: Both Sides | 8 | 7 | 6
  Improved: Either Side | 10 | 10 | 10

5. Secondary Outcome: Number of Participants With Satisfaction Responses as Assessed by Patient Satisfaction Questionnaire (PSQ) at Day 90 Post-treatment
Description: Participant satisfaction was determined by scores on PSQ completed at 90 days post-treatment. The participant completed this assessment while referring to baseline photos on a sponsor-supplied electronic tablet and a hand mirror. Participants were requested to provide information on "Please indicate what you think about how the treated areas of your lower face and neck look today. With your face relaxed (do not smile), look in the mirror at the treated area on both sides of your face and compare to the photos taken of both sides of your face prior to your study treatment." First questionnaire was as "Compared to when you started the study, how do your lower face, under your chin, and your upper neck look today?" Improved (much improved, improved, little improved), no change, worse. Second questionnaire was "How would you characterize your satisfaction with the treatment?" Satisfied (extremely satisfied, satisfied, slightly satisfied), neither satisfied or dissatisfied, dissatisfied.
Time Frame: Day 90
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
Number analyzed (Participants) | 21 | 19 | 16
Participants
  Improved | 18 | 15 | 16
  Satisfied | 17 | 13 | 14

ADVERSE EVENTS:
Time Frame: Baseline up to Day 90
Description: The investigator asked the participants for adverse events (AEs) systematically at each visit.
Arm/Group | Group EL 2: Ultherapy | Group EL 3: Ultherapy | Group EL 4: Ultherapy
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19 | 0/20
Other Adverse Events (participants affected / at risk) | 7/21 | 1/19 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group EL 2: Ultherapy (N=21) | Group EL 3: Ultherapy (N=19) | Group EL 4: Ultherapy (N=20)
Bruising/Ecchymosis (Injury, poisoning and procedural complications) | 3 | 0 | 1
Erythema/Redness (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Edema (Metabolism and nutrition disorders) | 2 | 0 | 0
Itching/Pruritus (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Tingling/Paresthesia/Numbness/ Nerve-related transient pain (Nervous system disorders) | 0 | 0 | 2
Nausea, Weakness (General disorders) | 0 | 0 | 1
Skin Pigmentation Change (Hypo-, Hyperpigmentation) (General disorders) | 0 | 1 | 0
Tenderness/Soreness/Pain/ Sensitivity to Touch (General disorders) | 1 | 0 | 0
Welting/Raised Areas of Edema (General disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2018-01-26): https://cdn.clinicaltrials.gov/large-docs/35/NCT03351335/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/35/NCT03351335/SAP_001.pdf